CLINICAL TRIAL: NCT02015299
Title: Off taRget Effects of Linagliptin monothErapy on Arterial Stiffness in Early Diabetes
Acronym: RELEASE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: dr. DJ Mulder (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor-Investigator, dr. DJ Mulder, MD, PhD, University Medical Center Groningen
Organization: University Medical Center Groningen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL43473.042.13
Record Dates: First submitted 2013-12-09; First posted 2013-12-19 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes; Pulse Wave Velocity; Dipeptidyl peptidase (DPP)-4 inhibitors; Linagliptin; Arterial Stiffness; Subclinical arterial inflammation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Linagliptin; Dipeptidyl-Peptidase IV Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Linagliptin (Experimental): Linagliptin 5 mg/day + lifestyle advise
  Interventions: Drug: Linagliptin
- Placebo (Placebo Comparator): Matching placebo + lifestyle advise
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Linagliptin — one tablet linagliptin 5 mg/day for 26 weeks
  Other Names: Trajenta; DPP-4 inhibitor
  Arms: Linagliptin
Drug: placebo — one tablet matching placebo/day for 26 weeks
  Arms: Placebo

SUMMARY:
Diabetes is associated with an increased risk for developing premature macrovascular complications. The process of irreversible subclinical damage to the vasculature already starts during its preceding stages. Dipeptidyl peptidase (DPP)-4 inhibitors have been shown to attenuate vascular damage in preclinical studies. Off-target effects on adipose tissue inflammation, liver steatosis and atherosclerotic plaques have been extensively documented in animal studies.

Based on these considerations the investigators hypothesize that early therapy with the DPP4 inhibitor linagliptin in subjects with treatment naive type 2 diabetes will lead to beneficial effects on arterial stiffness as measured by pulse wave velocity.

DETAILED DESCRIPTION:
Patients with type 2 diabetes mellitus (T2DM) are at increased risk for developing premature macrovascular complications. The process of irreversible subclinical damage to the vasculature already starts during its preceding stages. At diagnosis, patients with T2DM already have evidence of subclinical vascular damage. Recent trials have shown no benefit of glucose lowering therapy when started later in the course of the disease, implicating that early interventions could be more effective in preventing macrovascular complications. Dipeptidyl peptidase (DPP)-4 inhibitors are oral antidiabetic drugs that increase the action of the naturally gut hormone glucagon-like peptide-1 (GLP-1), leading to improvement of postprandial insulin secretion, without hypoglycaemia or weight gain. DPP4 inhibitors improve beta-cell function and insulin resistance. More importantly, off-target effects on adipose tissue inflammation, liver steatosis and atherosclerotic plaques have been extensively documented in animal studies. Furthermore, DDP4 inhibitors improve the cardiovascular risk profile in small clinical studies. Based on these considerations the investigators hypothesize that early therapy with the DPP4 inhibitor linagliptin in subjects with type 2 diabetes will lead to beneficial effects on arterial stiffness, blood pressure and inflammatory markers independent of its effects on glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age 30 to 70 years, AND
* Treatment naïve type 2 diabetes, as defined as t
* Fasting plasma glucose ≥ 7.0 mmol/l, OR
* Random plasma glucose ≥ 11.1 mmol/l, OR
* HbA1c ≥6,5%
* Written informed consent
* Assessable Pulse Wave Velocity measurement at screening

Exclusion Criteria:

* Current or previous use of glycemic control medications
* Type 1 diabetes
* Gestational diabetes mellitus
* Other specific types of diabetes due to other causes, e.g., genetic defects in β-cell function, genetic defects in insulin action, diseases of the exocrine pancreas (such as cystic fibrosis), and drug- or chemical-induced (such as in the treatment of HIV/AIDS or after organ transplantation)
* Uncontrolled hypertension, defined as systolic blood pressure >160 or a diastolic blood pressure >100 mmHg at screening visit
* Severe dyslipidemia indicating primary dyslipidemia, defined as total cholesterol >8 mmol/l, triglycerides >10 mmol/l of high density lipoprotein cholesterol <0.6 mmol/l
* Current use of weight loss medication or previous weight loss surgery
* History of severe gastrointestinal disease
* Clinical contraindications to DPP4-inhibitors
* Previous cardiovascular disease, defined as stable coronary artery disease or acute coronary syndrome, stroke or transient ischemic attack, peripheral artery disease
* Symptomatic heart failure, New York Heart Association (NYHA) class II-IV
* Women who are currently pregnant,planning to become pregnant,breastfeeding women, or women with child bearing potential not using appropriate contraceptive measures
* Clinically significant liver disease or hepatic function greater than 3 times upper limit of normal
* Known impaired renal function or eGFR <30 ml/min/1.73m2
* Patients who are mentally incompetent and cannot sign a Patient Informed Consent
* Current active malignancy or in the previous 6 months
* Documented HIV infection
* Use of rifampicin

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-03; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
change from baseline carotid-(right) femoral arterial Pulse Wave Velocity (PWV) at 26 weeks | baseline, week 26

SECONDARY OUTCOMES:
Secondary vascular study parameters | baseline, week 4, week 26, and 4 weeks after treatment discontinuation (week 30)
  * Central Blood Pressure (CBP) and Augmentation Index (AI) obtained from pulse wave analysis, using Sphygmocor
  * Carotid-(left) radial arterial PWV, using Sphygmocor
Subclinical vascular inflammation (FDG PET-CT) | 26 weeks
  Target-to-background ratios (TBRs) (18)F-fluorodeoxyglucose positron emission tomography computed tomography coregistration (FDG PET-CT)

OTHER OUTCOMES:
Body Mass Index and Waist-to-Hip ratio | baseline, week 4, week 26, and 4 weeks after treatment discontinuation (week 30)
  Body Mass Index and Waist-to-Hip ratio
Blood pressure | baseline, week 4, week 26, and 4 weeks after treatment discontinuation (week 30)
  24-hours ambulatory blood pressure measurement (24-ABPM)
Advanced glycation end products | baseline, week 4, week 26, and 4 weeks after treatment discontinuation (week 30)
  Skin AGE deposition measured and plasma levels of AGEs
plasma markers of inflammation | baseline, week 26
plasma markers of endothelial dysfunction | baseline, week 26
Glycemic indices | baseline, week 4, week 26, and 4 weeks after treatment discontinuation (week 30)
  Fasting glucose (FPG) and 2-hour post OGTT glucose (OGTT), HbA1c
albuminuria | baseline, week 4, week 26, and 4 weeks after treatment discontinuation (week 30)
  Urinary albumin/creatinine ratio
Lifestyle | baseline, week 26
  Intake of energy, Eating behaviour, and Physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Pieter W Kamphuisen, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Derived] Reijrink M, de Boer SA, Spoor DS, Lefrandt JD, Lambers Heerspink HJ, Boellaard R, Greuter MJ, Borra RJH, Hillebrands JL, Slart RHJA, Mulder DJ. Visceral adipose tissue volume is associated with premature atherosclerosis in early type 2 diabetes mellitus independent of traditional risk factors. Atherosclerosis. 2019 Nov;290:87-93. doi: 10.1016/j.atherosclerosis.2019.09.016. Epub 2019 Sep 25. PMID 31604171
- [Derived] de Boer SA, Hovinga-de Boer MC, Heerspink HJ, Lefrandt JD, van Roon AM, Lutgers HL, Glaudemans AW, Kamphuisen PW, Slart RH, Mulder DJ. Arterial Stiffness Is Positively Associated With 18F-fluorodeoxyglucose Positron Emission Tomography-Assessed Subclinical Vascular Inflammation in People With Early Type 2 Diabetes. Diabetes Care. 2016 Aug;39(8):1440-7. doi: 10.2337/dc16-0327. Epub 2016 Jun 8. PMID 27281773